CLINICAL TRIAL: NCT02701491
Title: Effect of Ginger on Nausea and Vomiting Related to Acute Gastroenteritis in Pediatric Age
Brief Title: Effect of Ginger on Nausea and Vomiting During Acute Gastroenteritis in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 273/15
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginger (Experimental): Ginger
  Interventions: Dietary Supplement: Ginger
- Placebo (Placebo Comparator): Placebo-no intervention
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger — ginger
  Arms: Ginger
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The acute gastroenteritis is a very common problem in children. The frequency and duration of this condition involves a high discomfort for the child and his family, and significant costs, in connection with the purchase of therapeutic aids, medical visits, days of work lost by parents, requiring hospitalization. Vomiting is a typical symptom of the majority of the cases of acute gastroenteritis and is very often the cause of failure of oral rehydration use and hospitalization.

To limit vomiting and facilitate oral rehydration have been proposed several pharmacological strategies. Unfortunately, these therapies are unsuccessful (domperidone), expensive and side effects (ondansetron and metoclopramide) and therefore contraindicated in patients of pediatric age.

The administration of some medicinal herbs is able to induce an effective anti-emetic power. Among the various types of plants studied, the rhizome of Zingiber officinale, commonly known as ginger is used as an antiemetic in various traditional systems of medicine for over 2000 years. There are several scientific evidence on the beneficial properties of ginger, including antioxidant, antimicrobial, anti-inflammatory and anti-allergic . It was also demonstrated that ginger is effective in resolving the post-operative nausea and vomiting and in pregnant. A recent meta-analysis has confirmed that ginger is effective in non-pharmacological treatment of nausea and vomiting in the early periods of pregnancy.

To date there are several formulations of the ginger on the market in Italy, and their use is fairly widespread in children for the treatment of vomiting by acute gastroenteritis in the absence of clinical evidence of efficacy.

The purpose of the proposed study is to demonstrate the effectiveness of treatment with ginger in reducing episodes of vomiting associated with acute gastroenteritis in children.

ELIGIBILITY:
Inclusion Criteria:

* Children, both sexes, aged 1-10 years,
* Diagnosis of acute gastroenteritis (duration less than 24 hours they had at least one episode of vomiting (no bile, no blood) in the previous four hours, with mild-state of dehydration moderate).

Exclusion Criteria:

* Children under 12 months of age and older than 10 years,
* concomitant presence of chronic diseases,
* malnutrition (z score for lower 3 standard deviations weight / height),
* severe dehydration,
* malformations of the gastrointestinal tract,
* malignancy,
* neurological diseases,
* metabolic diseases,
* eosinophilic esophagitis or other gastrointestinal diseases,
* history of functional dyspepsia or cyclic vomiting,
* history of abdominal surgery,
* history of food allergy ginger,
* renal failure and/or hypoalbuminemia

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in rate of subjects with persistence of symptoms | Change from baseline at 24 hours
  Rate of patients who present at least one more episode of vomiting following the beginning of the treatment assignment ( ginger or placebo) during the oral rehydration .

SECONDARY OUTCOMES:
Number of episodes of vomiting | Change from baseline at 24 hours
Change in rate of subjects with persistence of symptoms | Change from baseline at 48 hours
  Rate of patients who present at least one more episode of vomiting following the beginning of the treatment assignment ( ginger or placebo) during the oral rehydration .

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nocerino R, Cecere G, Micillo M, De Marco G, Ferri P, Russo M, Bedogni G, Berni Canani R. Efficacy of ginger as antiemetic in children with acute gastroenteritis: a randomised controlled trial. Aliment Pharmacol Ther. 2021 Jul;54(1):24-31. doi: 10.1111/apt.16404. Epub 2021 May 21. PMID 34018223